CLINICAL TRIAL: NCT03535805
Title: Randomized Trial of a Transdiagnostic, Cognitive and Behavioral Intervention Versus Treatment as Usual in School-aged Children With Emotional and Behavioral Disturbances
Brief Title: Transdiagnostic, Cognitive and Behavioral Intervention for in School-aged Children With Emotional and Behavioral Disturbances
Acronym: MindMyMind RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry); The Danish Mental Health Foundation (Other); Defactum, Central Denmark Region (Other Government)
Responsible Party: Principal Investigator, Pia Jeppesen, Ph.D., Senior Researcher, Specialist in Child and Adolescent Psychiatry, and Associate Professor, Institute for Clinical Medicine, Faculty of Health and Medical Sciences, University of Copenhagen, Denmark., Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The Mind My Mind Trial
Record Dates: First submitted 2018-04-30; First posted 2018-05-24 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Anxiety; Anxiety Disorders; Depressive Symptoms; Depressive Disorders; Problem Behavior; Oppositional Defiant Disorder; Conduct Disorder; Other Behavioral and Emotional Disorders With Onset Usually Occurring in Childhood and Adolescence
Keywords: Cognitive and Behavioral Therapies; Children and Adolescents; Community Health Care; Early Intervention
MeSH Terms: conditions — Anxiety Disorders; Depression; Depressive Disorder; Problem Behavior; Oppositional Defiant Disorder; Conduct Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The RCT is a parallel, two-arm, superiority trial comparing MMM with TAU for children aged 6-16 years with emotional and behavioural difficulties.
  This primary outcome is the parent-reported SDQ-impact of problems (range 0-10). The sample size calculation was based on the parameters from the feasibility RCT. Given an estimated standard variation (SD)=2.7, significance level=0.05, and power=0.90, the sample required to detect (or reject) a difference of at least 1.0 point is N=308. This sample size is also sufficient to detect clinically meaningful group differences in secondary outcome (e.g. 7.5% versus 16% reporting harm).
  The expected rate of attrition is 0.25. Hence, the investigators need to include 308/0.75=412 children to be randomly allocated (1:1). The central randomization uses concealed allocation sequences with variable block size, and stratification by region, age (6-10 or 11-16 years) and Top-problem (anxiety, depression, behavioural problems).
Who Masked: Outcomes Assessor
Masking Description: The statistical evaluation of the effects of MMM versus TAU will be carried out by researchers who will be masked for the treatment allocation.
  The central research-organization DEFACTUM is responsible for holding separate key files documenting the random allocation to treatment group and linking the ID numbers to the personal civil registration numbers. The analysts will be masked for treatment allocation until they have tested the primary and secondary hypotheses and confirmed or rejected the study hypotheses.
  It is not possible to mask the participants and the therapists in this study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind My Mind (MMM) (Experimental): Mind My Mind (MMM)
  Interventions: Behavioral: Mind My Mind (MMM)
- Treatment as Usual (TAU) (Active Comparator): Treatment as Usual (TAU)
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Mind My Mind (MMM) — Mind My Mind (MMM) is a new transdiagnostic and modular cognitive and behavioural therapy (CBT) program comprising evidence-based interventions for children and adolescents with anxiety, depression or disruptive behavior.
  MMM manual consists of evidence-based CBT methods that are organized into modules. The intervention is tailored to the individual child by the dosing and the sequencing of the modules. Trauma-focused CBT is available. Parents are engaged in child's therapy and support the child in doing the homework. Parent management training is offered for behavioral disturbances. The educational psychologists deliver the therapy after one-week training in the manual, followed by weekly supervision. The treatment fidelity is monitored by video observation of therapy sessions (>20%).
  The MMM training program consists of 9-13 sessions plus one booster, all completed within 17 weeks.
  Arms: Mind My Mind (MMM)
Behavioral: Treatment as Usual (TAU) — The parents in the TAU group are offered two sessions (week 2 and week 17) to support their attempts to seek help for the child in the municipality. This coordination is provided by psychologists (or other local professionals) who hold records of the currently available treatment options in the municipality. The TAU vary considerably from no intervention to counselling, talk therapy, pedagogical advice, network meetings, and/or individual support in the school setting. Some children are offered CBT interventions, but access to manualized treatment is generally very limited.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Background

Impairing emotional and behavioural problems are common in children and adolescents and mark a three-fold increased risk of mental disorder in young adulthood. Evidence-based psychological interventions are recommended for indicated prevention and first-line treatment, but access to treatment is often limited.

A new, modular cognitive and behavioural therapy program Mind My Mind (MMM) comprising evidence-based interventions for children with emotional and behavioral problems was designed to be delivered by educational psychologists in the Danish municipalities.

A feasibility RCT (NCT03448809), demonstrated that the study design was acceptable among children, parents, and therapists, and it provided data to estimate the sample size needed for the definitive RCT. The investigators test the hypothesis that the parent-reported impact of mental health problems will be significantly lower for children in the MMM group as compared with children in the TAU group after the 18-week intervention period (primary hypothesis), and after follow-up at week 26 (first secondary hypothesis).

Aim

To investigate the effects and cost-effectiveness of MMM compared with TAU for children and adolescents with impairing anxiety, depressive symptoms and/or behavioral problems. Both beneficial and harmful effects are evaluated.

Methods

The study compares the new modular MMM with TAU for children aged 6-16 years with anxiety, depressive symptoms or behavioral problems impacting on their daily and social life. The trial is conducted in four Danish municipalities in the period from September 2017 to April 2019. Participants are children with indicated needs.

The parents sign up the child for assessment in the Pedagogical Psychological Services in the Municipalities. The assessment includes web-based standardized questionnaires for child and parent: 1) the strengths and difficulties questionnaire (SDQ), 2) Spence Children's Anxiety Scale, 3) Mood and Feelings Questionnaire, and 4) family, social and school functioning. The questionnaires are supplemented with a clinical psychopathological interview by a trained psychologist. The investigators exclude children with 1) low levels of problems and no indicated needs, or 2) high levels of problems and need of referral to the Child and Adolescent Psychiatry.

412 children will be included and randomized (1:1) to MMM versus TAU. MMM is supported by a central organization, who is responsible for the education and weekly supervision of the therapists, and the web-based data collection and feedback of data in real time to therapists and researchers. All outcomes are self-, parent- and teacher-reported scores on standardized questionnaires administered at baseline, week 18 and week 26. At entry, the child and the parents own description of the Top-problem is recorded and scored on a 10-point likert scale. The Top-problem and impact of problem is scored by parent and child every second week during the intervention period, and the progress is monitored by the therapists in the MMM group. Information on costs is gathered through administrative registers and questionnaires at baseline, week 18, and week 26.

Primary objectives and outcome measures

This primary outcome is measured with the parent-reported SDQ impact-scale. The minimum relevant difference in impact of mental health problems was set at 1.0 corresponding to a change from severe to moderate, or from moderate to little-or-no impact in one of five domains of child's life: distress, home-life, friendships, classroom learning and leisure activities.

Secondary objectives and outcomes measures

The key secondary hypotheses are that the children in the MMM group will show significantly lower levels of parent-reported anxiety, depressive symptoms, functional impairment, Top-problems and behavioural problems, and better school attendance and quality-of-life as compared with the children in the TAU group at week 18.

All other outcomes are explored at week 18 and 26, including the primary and secondary measures of potential harm: 1) youths with severe and increased levels of self-reported suicidality, hopelessness and/or negative self-evaluation, and 2) youths with poor quality of life in relation to family, free time and friends.

Statistical analyses

All analyses will be intention-to-treat with two-sided significance tests. The investigators will use mixed models with repeated measures for continuous outcomes and generalized linear mixed model for binary and non-normally distributed outcomes. For the key secondary outcomes, the investigators will use the strategy of hierarchical testing allowing us to preserve the level of significance, α=0.05, as long as the null hypotheses are rejected. The incremental cost-effectiveness ratio will be calculated to analyze cost-effectiveness.

Perspectives

The results will guide policy makers in deciding whether to implement modular CBT-programs like the MMM.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6-16 years and in 0-9th grade (excluding the second semester of the 9th grade).
2. SDQ scores reported by the parent are above the lower cutoff: a total difficulties score of ≥14 and/or emotional problems ≥5, and/or conduct score ≥3; combined with a functional impairment score of ≥1. Scores above this cutoff place the child's difficulties within the top 10 percent of mental health problems in the general age-matched population in Denmark.
3. The child and parents determine one top problem that has to fall within the domains of anxiety, depressive symptoms or behavioral problems, according to the classification by the PPR (Pedagogical Psychological Services in the Municipalities) psychologist.
4. The child and at least one of the two parents understand and speak Danish sufficiently to participate in the treatment.
5. Written informed consent from the holders of the parental rights and responsibilities (usually both parents).

Exclusion Criteria:

1. Indications that the child may have a severe mental disorder like autism spectrum disorder, Attention Deficit Hyperactivity Disorder, schizophrenia-like psychosis, an eating disorder, severe obsessive-compulsive disorder, repeated self-harm, abuse or dependence of alcohol or psychoactive drugs or other mental disorder requiring referral to a more intensive assessment or treatment in child and adolescent mental health services (after systematic assessment and according to the usual recommendations and guidelines).
2. Indications of intellectual functional impairment, severe learning difficulties or other special needs that would interfere negatively with the MMM training. The judgment is made as a best estimate by the PPR psychologist on the basis of the available information. A formal intelligence test is not required.
3. A prior diagnosis of any developmental or mental disorder after assessment by the regional child and adolescent psychiatry, regardless of present status or treatment. A prior examination that did not result in a diagnosis of any specific mental health disorder will not exclude the child. The PPR psychologist must consult the PI who decides whether there is sufficient information to exclude the child because of a prior psychiatric history.
4. Prior participation in the MMM pilot or current study.
5. The child and/or parents are unable to participate in weekly sessions throughout the next 13-18 weeks.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 396 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
The child's impact of mental health problems reported by the parent on the Strengths and Difficulties Questionnaire (SDQ) | Week 0, 2, 4, 6, 8, 10, 12, 14, 18 and 26
  SDQ contains 25 items, each scored on a 3-point Likert scale (0, 1, 2), and divided into five sub-scales measuring emotional problems, behavioral problems, hyperactivity, peer problems and pro-social behavior. The total difficulties scale (range 0-40) sums up the difficulties across the first four problem areas.
  The extended version of the SDQ includes questions about child distress and interference of problems with home-life, friendships, classroom learning and leisure activities, and scores sum up the distress and the interference of problems on the impact scale (range 0-10).
  The minimum relevant difference in impact of mental health problems was set at 1.0 corresponding to a change from severe to moderate, or from moderate to little-or-no impact in one of the five domains of child's life.
  This primary outcome is measured with the parent-reported SDQ impact-scale (range 0-10) and analyzed in a mixed model with repeated measures adjusting for the stratification variables.

SECONDARY OUTCOMES:
Child' anxiety reported by the parent on 'Spence Children's Anxiety Scale (SCAS) | Week 0, 18 and 26
  The parent-reported SCAS comprises 38 items, rated on a four-point scale (0-1-2-3). The six subscales cover social phobia (SoP; six items), panic disorder and agoraphobia (Panic; nine items), generalized anxiety disorder (GAD; six items), obsessive-compulsive disorder (OCD; six items), separation anxiety disorder (SAD; six items) and fear of physical injury (Fear; five items). Each subscale is scored separately and added together for a total score reflecting overall anxiety symptoms. A validation of the Danish version of the SCAS in children and adolescents aged 7-17 years found good psychometric properties.
Child's depressive symptoms reported by the parent on the Mood and Feelings Questionnaire (MFQ) | Week 0, 18 and 26
  The parent-reported MFQ comprises 34 items, each rated on a three-point scale (0-1-2).
  The MFQ have well-established predictive validity for detection of depressive states and suicidality in epidemiological and clinical samples of children and adolescents aged 8-17 years, and the parent-reported MFQ has also demonstrated sensitivity for change with treatment.
Weiss Functional impairment rating Scale (WFIRS) | Week 0, 18 and 26
  The Weiss Functional Impairment Rating Scale-Parent Report (WFIRS) was designed to evaluate to what degree a child's behavior or emotional problems impacted on various domains of daily functioning. The questionnaire comprises 50 items, each rated on a four-point scale (0-1-2-3). Although it has only been validated (and found very sensitive for change) in clinical samples of children with ADHD, it focuses on the impact of emotional and behavioral problems in children. The six domains (subscales) cover: Family and home life, School and learning, Life skills, Self-Concept, Social activities, and Risk behaviors.
  Only the parent-reported version was used in the present study.
The self-reported physical and psychological well-being (two subscales from the KIDSCREEN). | Week 0, 18 and 26
  The KIDSCREEN is a Health-Related Quality of Life (HRQOL) questionnaire for children and adolescents aged from 8 to 18 years.
  It comprises parent- and youth-reported questionnaires. The investigators used the version with 27 items (rated on a five point scale, 1-2-3-4-5), containing five dimensions (subscales): Physical Well-Being, Psychological Well-Being, Autonomy & Parents, Peers & Social Support and School Environment.
  For the key secondary outcomes, the investigators use only the two self-reported subscales: 'Physical Well-Being' and 'Psychological Well-Being'.
The child's behavioural problems, reported by the parent on the Eyberg Child Behaviour Inventory (ECBI) | Week 0, 18 and 26
  The ECBI is a brief, parent-reported behavioral rating scale of externalizing problems in children of age 2-16 years. It consists of 36 items that assess typical problem behavior in children with oppositional and conduct disorders. Each item is rated on a 7-point Intensity Scale indicating how often the behaviors currently occur (0=Never, 4=sometimes, 7=always); and a Problem scale that identifies whether the child's behavior is problematic or not for the parent (1=yes, 0=no). Hence, the sum of scores on the 'Intensity Scale' measures the overall intensity of problem behavior, while the sum of scores on the 'Problem scale' measures the number of problematic behaviors.
Total emotional and behavioural difficulties, reported by parents (SDQ) | Week 0, 18 and 26.
  The SDQ total difficulties scale (range 0-40) sums up the difficulties across the four problem areas: emotional problems, behavioral problems, hyperactivity, and peer problems.
School attendance | Week 18 and 26
  The parent reports the frequency of days with school attendance problems within the last four weeks: 1) days with late attendance, 2) days not attending school with parental accept or knowledge, 3) days not attending school without parental knowledge (best estimate in retrospect)
Top-problem scores, parent-reported | Week 0, 2, 4, 6, 8, 10, 12, 14, 18 and 26
  At entry, the child and the parents own description of the Top-problem is recorded and scored on a 10-point likert scale (range 1-10).
  The Top-problem is scored by the parent during the intervention period in both treatment groups.
  The therapists monitor the scores in MMM training group.
The self-reported impact of mental health problems (SDQ, only children of age ≥ 11 years) | Week 0, 2, 4, 6, 8, 10, 12, 14, 18 and 26
  The SDQ impact scale (range 0-10) covering child distress and interference of problems with home-life, friendships, classroom learning and leisure activities.
  The impact scale is administered as part of the SDQ at week 0, 18 and 26; and as part of the new session-by-session questionnaire at week 2, 4, 6, 8, 10, 12, and 14.
The teacher-reported impact of mental health problems (SDQ) | Week 0, 18 and 26
  The teacher-reported version of the SDQ impact scale (range 0-6) covers child distress and interference of problems with friendships and classroom learning.
Self-reported anxiety reported (SCAS, only children of age ≥ 8 years) | Week 0, 18 and 26
  The parent-reported SCAS comprises 44 items, rated on a four-point scale (0-1-2-3). The self-reported version is longer than the parent-reported, because it includes six positive filler items.
Self-reported depressive symptoms (MFQ, only children of age ≥ 8 years) | Week 0, 18 and 26
  The parent-reported MFQ comprises 33 items, each rated on a three-point scale (0-1-2).
Self-reported Top-problem scores | Week 0, 2, 4, 6, 8, 10, 12, 14, 18 and 26
  The Top-problem is scored by the child during the intervention period in both treatment groups.
  The therapists monitor the scores in MMM training group.
The parent-reported Health-Related Quality of Life (HRQOL) of their child (KIDSCREEN) | Week 0, 18 and 26
  For other secondary outcomes, the investigators use all the parent-reported subscales of the KIDSCREEN: Physical Well-Being, Psychological Well-Being, Autonomy & Parents, Peers & Social Support and School Environment.
Self-reported emotional and behavioural difficulties (SDQ, only children of age ≥ 11 years) | Week 0, 18 and 26
  The SDQ total difficulties scale (range 0-40) sums up the difficulties across the four problem areas: emotional problems, behavioral problems, hyperactivity, and peer problems.
Teacher-reported emotional and behavioural difficulties (SDQ) | Week 0, 18 and 26
  The SDQ total difficulties scale (range 0-40) sums up the difficulties across the four problem areas: emotional problems, behavioral problems, hyperactivity, and peer problems.
Parental Stress Scale (PSS) | Week 0, 18 and 26
  The PSS is a parent-reported questionnaire with 18 items, each rated on a five point scale (0-1-2-3-4). It measures the stress a parent may experience in their role-function as parent.
The parent-reported Experience of Service Questionnaire (ESQ) | Week 18 and 26
  The parent-reported ESQ comprises seven items, each rated on a three-point scale (0-1-2). The Danish version was adapted from a longer English questionnaire asking young people and their parents how they felt about the psychiatric service they received. The brief Danish version proved useful in a recent study of efficacy of the Cool Kids program in Denmark.
The self-reported Experience of Service Questionnaire (ESQ) | Week 18 and 26
  The child-reported ESQ comprises seven items, each rated on a three-point scale (0-1-2).
The parent- and child-reported Child Health Utility 9D (CHU9D) | Week 0, 18 and 26
  CHU9D is a generic preference-based measure of health-related quality of life. It contains nine items, each with five response categories that assess the child's functioning across domains of worry, sadness, pain, tiredness, annoyance, school, sleep, daily routine and activities.
Parents' absence from work | Week 0, 18 and 26
  The parent reports the frequency of hours/days each of the parents have been absence from work within the last four weeks due to the problems of the child.
Treatment and support received by the child and the family | Week 0, 18 and 26
  The parent reports any support or treatment received by the child and/or family from the municipality, general practitioner, and private actors.
The primary measures of potential harms | Week 18 and 26
  Selected items from the Mood and Feelings questionnaire (MFQ), covering the last two weeks, and scored by the child: four items on Suicidality ("I thought that life wasn't worth living", "thoughts about death or dying", "I thought my family would be better off without me", "I thought about killing myself"), and four items covering Negative cognitions about guilt, hopelessness and self-evaluation ("I blamed myself for things that weren't my fault", "I thought there was nothing good for me in the future", "I hated myself", "I felt I was a bad person").
  If at least one out of the four items are scored "always" (the most severe response) at follow-up, but not at entry, then a potential harm is counted present (yes/no) in the domain of Suicidality and/or Negative cognitions.
The secondary measures of potential harm | Week 18 and 26
  Selected items from the KIDSCREEN covering the last week and scored by the child: five items on family relations/ free time ("Have you had enough time for yourself?", "Have you been able to do the things that you want to do in your free time?", "Have your parents had enough time for you?", "Have your parents treated you fairly?", "Have you been able talk to your parents when you wanted to?"; and four items on friends ("Have you spent time with your friends?", "Have you had fun with your friends?", "Have you and your friends helped each other?", "Have you been able to rely on your friends?").
  If at least one out of the five and four items, respectively, are scored "always" (the most severe response) at follow-up, but not at entry, then a potential harm is counted present (yes/no) in the domain of family relations/free time and/or friends.
Costs | Week 26
  Costs of the Mind My Mind intervention and treatment as usual will be estimated.
Incremental cost-effectiveness ratio (ICER) | Week 26
  The ICER using the primary outcome SDQ impact score as effect measure will be calculated (CEA) as well as the ICER using quality-adjusted life years, derived from the CHU9D score, as effect measure (CUA).

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jeppesen, PhD, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Mental Health Services in the Capital Region, Denmark, Copenhagen, Denmark

REFERENCES:
- [Derived] Rimvall MK, Vassard D, Nielsen SM, Wolf RT, Plessen KJ, Bilenberg N, Thomsen PH, Thastum M, Neumer SP, Puggaard LB, Pedersen MMA, Pagsberg AK, Silverman WK, Correll CU, Christensen R, Jeppesen P. Effect modification of an effective transdiagnostic cognitive behavioral psychotherapy in youths with common mental health problems: Secondary analyses of the randomized mind-my-mind trial. Eur Neuropsychopharmacol. 2023 Sep;74:64-75. doi: 10.1016/j.euroneuro.2023.05.004. Epub 2023 Jun 4. PMID 37279641
- [Derived] Jeppesen P, Wolf RT, Nielsen SM, Christensen R, Plessen KJ, Bilenberg N, Thomsen PH, Thastum M, Neumer SP, Puggaard LB, Agner Pedersen MM, Pagsberg AK, Silverman WK, Correll CU. Effectiveness of Transdiagnostic Cognitive-Behavioral Psychotherapy Compared With Management as Usual for Youth With Common Mental Health Problems: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Mar 1;78(3):250-260. doi: 10.1001/jamapsychiatry.2020.4045. PMID 33355633

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03535805/SAP_000.pdf
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT03535805/Prot_001.pdf